CLINICAL TRIAL: NCT01599273
Title: Treatment of Upper Eyelid Retraction Related to Thyroid-associated Ophthalmopathy Using Subconjunctival Triamcinolone Injections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2012-0164
Record Dates: First submitted 2012-05-10; First posted 2012-05-16 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Thyroid-associated Ophthalmopathy
Keywords: thyroid-associated ophthalmopathy; triamcinolone; retraction; swelling
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triam inj (Experimental)
  Interventions: Drug: subconjunctival triamcinolone injection
- observation group (No Intervention)

INTERVENTIONS:
Drug: subconjunctival triamcinolone injection — Patients are randomized into two groups: Injection (Group 1) and observation-only controls (Group II). In Group I, patients were treated with 1-3 injections of 20 mg triamcinolone acetate using a 30-gauge needle into the subconjunctival region of the lid between the conjunctiva and Muller's muscle. Injections were stopped after 1-2 injections if both swelling and retraction resolved completely, or if one eye scored 0 and the contralateral eye scored 1, and there existed no patient concern after physician inquiry regarding function and cosmetic appearance.
  Arms: Triam inj

SUMMARY:
Thyroid-associated ophthalmopathy (TAO) is an autoimmune process that can affect the orbital and periorbital tissues and the thyroid gland. Periorbital inflammation can cause swelling, fatty infiltration, and scarring of the eyelid muscles resulting in eyelid retraction and upper scleral exposure, which is the most common clinical features of TAO.Even with mild eyelid retraction and swelling, most patients become disappointed and depressed due to their cosmetically unacceptable appearance, and they are unwilling to wait for spontaneous resolution or a clinically inactive period for surgical intervention. Thus, most ophthalmologists and endocrinologists recommend surgery in the chronic burnt-out stage. Several treatment options have been described for correction of eyelid retraction, including Botox and filler injection, and surgeries in the burnt-out stage such as lowering the upper lid by recessing the levator muscle, excision of Müller's muscle, introducing a spacer, or myotomies.Surgical options have significant risks as well as an unpredictable course and outcome in some cases. Several authors have reported that subconjunctival botulinum toxin injection provides an immediate, effective treatment by reducing excessive levator function in patients who suffer from disfiguring eyelid appearance and do not want to wait for surgery for upper eyelid retraction.Botox treatment is usually temporary. However, unwanted ptosis, although temporary, was observed in five out of 24 patients (20.8%) in the study by Costa, which may be even more disappointing and cosmetically unacceptable to some patients.Recently, hyaluronic acid gel fillers, which were injected into the subconjunctival levator-Muller plane, demonstrated efficacy in managing Graves' eyelid retraction in three patients.However, complications such as a lumps, fluid buildup, and skin pigment darkening may occur using this technique.Steroid treatment represents a well-established TAO management strategy due to its anti-inflammatory and immunosuppressive actions. However, multiple systemic side effects such as diabetes, infection, hypertension, osteoporosis, and stomach ulcers are major drawbacks of systemic steroid treatment. Due to limitations of systemic steroid treatment, several studies reported TAO improvement with periorbital injections of methylprednisolone and triamcinolone, primarily focusing on reducing proptosis and diplopia. So far, however, only a single small case series study has suggested that an injection of 20 mg triamcinolone into the subconjunctival region of the lid, between the conjunctiva and Muller's muscle, improves upper eyelid retraction within 1 month in three of the four patients. The investigators are not aware of any study designed to demonstrate the treatment efficacy of locally administered triamcinolone to improve eyelid retraction and swelling in a prospective manner. Therefore, we aimed to evaluate both the short-term and long-term effects of subconjunctival triamcinolone injections in treating eyelid retraction and inflammatory swelling caused by TAO.

ELIGIBILITY:
Inclusion Criteria:

* TAO symptom duration less than 6 months
* Eyelid retraction or swelling
* Participants who is able to sign a consent agreement and proceed study

Exclusion Criteria:

* Previous steroid or radiation treatment for TAO
* Compressive optic neuropathy
* Suspicious of glaucoma or high risk of intraocular pressure elevation
* Patients with eyeball pain and/ or 4 or more of Mourtis' clinical activity score(CAS)
* Patients who are not in euthyroid status at the start of study period and or the whole duration of study period
* Pregnant or breast feeding women

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
change of Eyelid retraction grade | At 3, 6, and 9 weeks after the initial injection, and finally at 24 weeks post-injection.
  Injection (Group 1) and observation-only controls (Group II). At 3, 6, and 9 weeks after the initial injection, and finally at 24 weeks post-injection for group I. In Group II, eyelids were evaluated at 9 and 24 weeks after the initial visit.

SECONDARY OUTCOMES:
change of Eyelid swelling | At 3, 6, and 9 weeks after the initial injection, and finally at 24 weeks post-injection
  Patients are randomized into two groups: Injection (Group 1) and observation-only controls (Group II). At 3, 6, and 9 weeks after the initial injection, and finally at 24 weeks post-injection. In Group II, eyelids were evaluated at 9 and 24 weeks after the initial visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Lee SJ, Rim TH, Jang SY, Kim CY, Shin DY, Lee EJ, Lee SY, Yoon JS. Treatment of upper eyelid retraction related to thyroid-associated ophthalmopathy using subconjunctival triamcinolone injections. Graefes Arch Clin Exp Ophthalmol. 2013 Jan;251(1):261-70. doi: 10.1007/s00417-012-2153-y. Epub 2012 Sep 12. PMID 22968823